CLINICAL TRIAL: NCT01962389
Title: First in Human Study of Winsor Laser Catheter
Brief Title: First in Human Study of Winsor Laser Catheter: A Prospective Registry to Evaluate The Safety and Performance of the Winsor Laser Catheter in the Treatment of In-Stent Restenosis
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Spectranetics Corporation (Industry)
Collaborators: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Winsor - 001
Record Dates: First submitted 2013-10-07; First posted 2013-10-14 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Femoropopliteal In-Stent Restenosis
Keywords: ISR, Laser, SFA, PAD

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Winsor Laser Catheter (Experimental)
  Interventions: Device: Winsor Laser Catheter

INTERVENTIONS:
Device: Winsor Laser Catheter

SUMMARY:
The study will evaluate the procedural safety and efficacy of the Winsor Laser Catheters for the treatment of In-Stent Restenosis (ISR) in the Superficial Femoral Artery (SFA)

ELIGIBILITY:
Inclusion Criteria:

1. Patient age ≥ 18 years.
2. Rutherford Category 2-4.
3. Subject has been informed of the nature of the study, agrees to participate and has signed an Ethics Committee approved informed consent form.
4. Documentation of significant ISR defined as >50% stenosis and >5 cm in length determined by diagnostic angiogram or duplex ultrasound.
5. A previously deployed bare nitinol stent(s) in the femoropopliteal segment extending from the ostium of the SFA to 1 cm above the tibioperoneal trunk. A guidewire has successfully traversed the target treatment segment, or is able to cross using standard support catheter crossing techniques, is angiographically documented to be within true lumen and not placed through stent struts. Guidewire access may obtained via contralateral, ipsilateral or retrograde approach. If a retrograde guidewire approach is used to cross the target lesion, guidewire exchange and an antegrade approach is required prior to treatment with the Winsor Laser Catheter.
6. One or more patent tibial vessel(s) defined as <50% stenosis thoughout the segment with outflow to the foot.
7. Successful treatment of any inflow lesion(s) defined as final residual stenosis <30%.

Exclusion Criteria:

1. Patient is pregnant.
2. Has known uncontrollable hypercoagulable condition, or refuses blood transfusion.
3. Any co-morbid condition that in the judgment of the physician precludes safe percutaneous intervention.
4. Crossing devices other than guidewire support catheters.
5. Type 4 or 5 stent fracture as assessed by angiography.
6. Target lesion is located within a covered stent.
7. Acute limb ischemia

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoint | up to 48 hours
  Freedom from Major Adverse Events (MAE) through hospital discharge:
  * All-cause peri-procedural death
  * Target limb amputation (above or below the ankle)
  * Target limb re-intervention
  * Target limb-related death

SECONDARY OUTCOMES:
Efficacy | During Interventional Procedure
  Procedural success defined as the percent of target lesions that achieve ≤30% residual stenosis at the completion of the procedure (laser atherectomy and any adjunctive treatment) as determined by an independent angiographic core lab.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Mena, MD, Principal Investigator — Yale University
Locations (1):
- Centro Cardiovascular Colombiano, Medellín, Colombia